CLINICAL TRIAL: NCT05728996
Title: Netherlands Cohort Study on Acute HIV Infection
Acronym: NOVA
Status: Recruiting | Type: Observational
Sponsor: Prof. Jan Prins (Other)
Collaborators: UMC Utrecht (Other); Rijnstate Hospital (Other); Erasmus Medical Center (Other); Onze Lieve Vrouwe Gasthuis (Other); Radboud University Medical Center (Other); Maasstad Hospital (Other); DC Clinics (Unknown); Amsterdam UMC, location VUmc (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Prof. Jan Prins, Full professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: NL51613.018.14
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Acute HIV Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum PBMC Leukapheresis GALT Lymph node Cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: "standard": only routine diagnostic procedures are performed
- Group 2A: "less invasive": in addition to routine monitoring, patients also undergo semen sampling
- Group 2B: "less invasive": in addition to routine monitoring, patients undergo semen sampling and/or leukapheresis.
- Group 3: "extended": patients undergo (in addition to routine sampling) semen sampling, invasive tissue sampling (GALT and/or lumbar puncture) and leukapheresis.

SUMMARY:
Investigation of the size, variability and localization of the (pro) viral reservoir and the properties of HIV-specific immune response related to "post-treatment viral remission' achievement and / or duration. In addition we will study the factors that determine latency in the different host cells, their sensitivity to induction of replication competent virus by various agents and the potential application of these agents in "post-treatment viral remission".

This all will be studied in patients included during acute phase of the infection who start antiretroviral therapy immediately upon diagnosis.

DETAILED DESCRIPTION:
Rationale: There is renewed interest in finding a cure for HIV infection. Recent studies show that in a select group of individuals the initiation of combination anti-retroviral therapy (cART) during the early phase of infection results in long-term absence of viremia following treatment interruption after prolonged treatment. These patients are described as having achieved a "post-treatment viral remission". There are many unsolved issues regarding the question which virological and immunological factors determine which individuals achieve a "post-treatment viral remission". First studies suggest that the early reduction of viral reservoir size and potential accompanying preservation of immune function may be important factors. Furthermore, patients that initiate cART during acute infection are potential candidates for additional therapeutic strategies, such as latency reversing agents (LRAs) or therapeutic vaccination.

Objectives: The primary objective of the NOVA study is the establishment of a prospective cohort study of patients that initiate cART during the acute infection phase, aiming at achieving "post-treatment viral remission". The secondary objective is to characterize the viro-immunological factors that correlate with achievement of "post-treatment viral remission" for several years in these patients.

Study design: Prospective cohort study. Study population: The study population includes patients diagnosed with an AHI (Fiebig stage I-V, 20 in each stage). As a control group only for comparison of the lymph node viral reservoir and immune responses after 3 years of cART, 20 age-matched patients will be included who start cART in the chronic phase of infection. This control group is recruited to provide PBMCs and a LN sample for comparison purposes. Patients will be recruited over a period of 5 consecutive years.

Intervention: Patients diagnosed with an acute HIV infection (AHI) are offered immediate standard first-line cART. In consenting patients, at several time points samples will be obtained to analyze the size and characteristics of the viral reservoir and the accompanying immune function. Three groups are assembled based on the preparedness of individual patients to participate in the extensiveness of sampling. Patients that accept early treatment and follow-up but decline additional blood and tissue sampling (lymph node, GALT and cerebral spinal fluid (CSF)) are included in group 1 ("standard") and only routine diagnostic procedures are performed. Patients willing to undergo, in addition to routine monitoring, leukapheresis, semen and blood sampling for PBMC and virological analyses are included in group 2 ("less-invasive"). In group 3 ("extended") additional tissue and CSF sampling will be performed for the proposed viro-immunological analyses.

Main study parameters / endpoints: We will investigate the size, variability and localization of the (pro) viral reservoir and the properties of HIV-specific immune response and relate these to "post-treatment viral remission' achievement and / or duration. In addition we will study the factors that determine latency in the different host cells, their sensitivity to induction of replication competent virus by various agents and the potential application of these agents in "post-treatment viral remission".

This set up allows to guide the duration of cART based on viro-immunological parameters and to adjust cART in case better cART strategies may become available in the future. Furthermore, based on the available data that show preservation of immunity and reduction in viral reservoir size, the AHI patients that start therapy early may have better responses to future cure strategies such as therapeutic vaccination or LRAs.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Offering treatment in early HIV infection is currently recommended in clinical guidelines for treatment of HIV infection 1. This recommendation is based on studies showing improvement of markers of disease progression 2;3 decrease of severity of acute disease, lowering of the viral setpoint (associated with disease progression) 4;5;6 and a reduction in size of the viral reservoir 7. The burden and risks associated with study participation are related to tissue sampling: lymph node excision biopsies, sigmoid biopsies and lumbar puncture at three and leukapheresis at two timepoints during the study (week 0 (baseline), week 24 and 3 years). The risks of sampling are considered minimal (see also section on "sampling"). Furthermore, since potential discontinuation of cART in future can only be guided by size of (tissue) viral reservoir, the sampling is considered to be necessary for treatment guidance. In order to minimize burden associated with study visits, we aim to combine visits for routine clinical care with routine clinical visits.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to store samples and perform genetic testing.
* Separate written informed consent for invasive sampling procedures: leukapheresis, sigmoidoscopy with biopsies, lymph node excision biopsy and lumbar puncture, with storage of samples.
* Age >= 18 years
* An acute HIV-1 infection, defined according to the Fiebig stages I-IV (acute infection), as described in the previous paragraph (HIV-1 RNA positive and 4th generation ELISA negative or HIV-1 RNA positive and 4th generation HIV ELISA positive with indeterminate Western Blot). Patients in Fiebig stage V and VI (recent infection) will only be included if they have a documented negative HIV test 6 months prior to the positive test or if they are in Fiebig stage V with a p31 negative blot
* Female subjects should be willing to use adequate contraception.

Exclusion Criteria:

* Contraindication for proposed cART regimen (e.g. impaired renal function).
* Mental disorder that in the view of the investigator would interfere with adherence to the treatment or the study procedures, or the decision to participate in the study.
* Immunosuppressive medication or other diseases associated with immunodeficiency.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes patients diagnosed with an AHI (Fiebig stage I-V, 20 in each stage). As a control group only for comparison of the lymph node viral reservoir and immune responses after 3 years of cART, 20 age-matched patients will be included who start cART in the chronic phase of infection. This control group is recruited to provide PBMCs and a LN sample for comparison purposes. Patients will be recruited over a period of 5 consecutive years.
Sampling Method: Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
The establishment of a prospective cohort study of patients that initiate cART during the acute infection phase, aiming at achieving "post-treatment viral remission". | 10 years

SECONDARY OUTCOMES:
Characterize the viro-immunological factors that correlate with achievement of "post-treatment viral remission" for several years in these patients. | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Paassen P, Dijkstra M, Peay HL, Rokx C, Verbon A, Reiss P, Prins JM, Henderson GE, Rennie S, Nieuwkerk PT, de Bree GJ. Perceptions of Rapid Antiretroviral Therapy Initiation Among Participants of The Netherlands Cohort Study on Acute HIV Infection. AIDS Res Hum Retroviruses. 2024 May;40(5):286-292. doi: 10.1089/AID.2022.0169. Epub 2023 Oct 30. PMID 37791419